CLINICAL TRIAL: NCT04886011
Title: Evaluation of Novel Topical Camel Whey Protein Gel for the Treatment of Recurrent Aphthous Stomatitis: Randomised Clinical Study
Brief Title: Camel Whey Protein Gel for the Treatment of Aphthous Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Principle investivagor and lecturer of oral medicine and periodontology, faculty of dentistry, kafrelsheikh university, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFSAPH2021
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Aphthous Stomatitis, Recurrent; Antioxidative Stress
MeSH Terms: conditions — Sutton disease 2

STUDY DESIGN:
Intervention Model Description: Methylcellulose gel
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo gel (Placebo Comparator): Methylcellulose gel was applied to the ulcer till complete healing
  Interventions: Combination Product: placebo gel
- camel whey protein gel (Experimental): camel whey protein dissolved in methycellulose gel was applied to the ulcer till complete healing
  Interventions: Combination Product: camel whey protein gel

INTERVENTIONS:
Combination Product: placebo gel — just methyl cellulose gel was applied to the ulcer
  Arms: placebo gel
Combination Product: camel whey protein gel — camel whey protein gel was prepared and dissolved in methyl cellulose gel base and applied to the ulcer
  Arms: camel whey protein gel

SUMMARY:
Higher prevalence of recurrent aphthous ulcer in young adults and the severity decreased with increasing age. The etiology of aphthous ulcer remains unclear. Other possible factors include trauma, drug use, deficiency in vitamin B12, folic acid, iron, stress, hormonal changes and metabolic diseases. Many topical agents such as local and systemic an- tibiotics, local antiseptics, topical NSAIDs, and topical corticosteroids are generally prescribed for symptomatic relief. Several approved drug for- mulations such as pills, mouthwash, sprays and paste such as vitamin B12, chlorhexidine mouthwash, steroid lozenges and local anesthetics are primarily suggested for the treatment of aphthous ulcer.

Camel whey protein gel was fabricated to get benefits of its antiinflammatory, immunomodulator, Antibacterial and antioxidant effects.

DETAILED DESCRIPTION:
40 cases of recurrent aphthous ulcer patients as the research object,were randomly divide into the study group and the control group, each with 20 cases of both sexes with age ranging from 18 years to 50 years.

Inclusion criteria consisted of the following: (a) clinical examination and confirmed history of recurrent oral ulcer, (b) recurrence of the oral ulceration, and (c) patients in good condition with no serious systemic disease. Eligible persons were excluded if they were administered antibiotics or glucocorticoids or accepted periodontal or dental treat- ments that interfered with the results of our experimental drugs.

the control group will be subjected to placebo gel consisting of methyl cellulose gel whereas the study group will use camel whey protein dissolved in methyl cellulose gel base. the gel will be applied 1 day after ulcer appearance and will be stopped after ulcer disappearance

ELIGIBILITY:
Inclusion Criteria:

* clinical examination and confirmed history of recurrent oral ulcer,
* recurrence of the oral ulceration
* patients in good condition with no serious systemic disease.

Exclusion Criteria:

* if they were administered antibiotics or glucocorticoids
* accepted periodontal or dental treat-ments that interfered with the results of our experimental drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
pain level | 1 week
  visual analog scale to measure pain level from 0 to 10. 0 means no pain at all and 10 means the most sever pain
ulcer duration | 10 days
  time extended from ulcer presence till disseverance

SECONDARY OUTCOMES:
immunological analysis | 10 days
  the values of serum TNF-α, Il1, IL6 were measured before and after gel application using flow cytometry

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - oral medicine and periodontology outpatient clinic, faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh
  - Walid Elamrousy, Kafr ash Shaykh

IPD SHARING:
Plan to Share IPD: No